CLINICAL TRIAL: NCT02647424
Title: A Comparison of Hormonal Profile and the Follicular Development Between Letrozole and Clomifene Citrate in Anovulatory Women With Polycystic Ovary Syndrome and Ovulatory Women
Brief Title: A Comparison of Letrozole and Clomifene Citrate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKU-VL-LCC
Record Dates: First submitted 2015-12-29; First posted 2016-01-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Polycystic Ovarian Syndrome; Subfertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCOS group (Other): PCOS women with anovulation
  Interventions: Drug: Letrozole; Drug: Clomiphene
- Ovulatory group (Other): Ovulatory group planned for intra-uterine insemination
  Interventions: Drug: Letrozole; Drug: Clomiphene

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg daily from Day 2 to 6
  Other Names: Letrozole group
Drug: Clomiphene — After one month of washout period, clomiphene 50 mg daily from day 2 to day 6 given
  Other Names: Clomiphene group

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrinopathies, affecting 5% to 10% of women of reproductive age. Women with PCOS suffer from anovulatory infertility. Following lifestyle modification with weight reduction in obese PCOS women, clomifene citrate (CC) is considered the first line treatment for ovulation induction (OI) in these women. 75-80% of women will ovulate after CC administration. However, there is a discrepancy between the ovulation rate and pregnancy rate, which was reported to be 22% per each ovulating cycles after CC. Other alternatives, including gonadotropin injections and laparoscopic ovarian drilling, carried different disadvantages, such as costly treatment and risks of ovarian hyperstimulation syndrome and multiple pregnancy rate in gonadotrophin therapy and surgical risks and risk of ovarian failure in surgical treatment.

The use of aromatase inhibitor, letrozole (LTZ), in reproductive medicine started in 2001. After this publication, there have been many groups of investigators studying the use of LTZ either in OI or ovarian stimulation in IVF cycles. A large multicentre randomized trial reported a significantly higher ovulation rate and live-birth rate comparing LTZ with CC. In majority of the publications, the multiple pregnancy rate was lower in LTZ group than in CC group. This can be attributed to the higher chance of monofollicular development after LTZ compared with CC. However, there is no information comparing the hormonal profile and follicular development after letrozole and CC.

Mild ovarian stimulation using LTZ or CC in conjunction with intrauterine insemination is commonly offered to ovulatory women with unexplained infertility, minimal endometriosis or mild factor to improve the pregnancy rate. There is again no information comparing the hormonal profile and follicular development after letrozole and CC in ovulatory women.

The aim of this study is to compare the hormonal profile after the use of LTZ and CC in anovulatory PCOS women and ovulatory women with unexplained subfertility. The hypothesis is that the FSH risk after LTZ is shorter than that of CC.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is one of the most common endocrinopathies, affecting 5% to 10% of women of reproductive age. Women with PCOS suffer from anovulatory infertility. Following lifestyle modification with weight reduction in obese PCOS women, clomifene citrate (CC) is considered the first line treatment for ovulation induction (OI) in these women. 75-80% of women will ovulate after CC administration. However, there is a discrepancy between the ovulation rate and pregnancy rate, which was reported to be 22% per each ovulating cycles after CC. Other alternatives, including gonadotropin injections and laparoscopic ovarian drilling, carried different disadvantages, such as costly treatment and risks of ovarian hyperstimulation syndrome and multiple pregnancy rate in gonadotrophin therapy and surgical risks and risk of ovarian failure in surgical treatment.

The use of aromatase inhibitor, letrozole (LTZ), in reproductive medicine started in 2001. After this publication, there have been many groups of investigators studying the use of LTZ either in OI or ovarian stimulation in IVF cycles. A large multicentre randomized trial reported a significantly higher ovulation rate and live-birth rate comparing LTZ with CC. In majority of the publications, the multiple pregnancy rate was lower in LTZ group than in CC group. This can be attributed to the higher chance of monofollicular development after LTZ compared with CC. However, there is no information comparing the hormonal profile and follicular development after letrozole and CC.

Mild ovarian stimulation using LTZ or CC in conjunction with intrauterine insemination is commonly offered to ovulatory women with unexplained infertility, minimal endometriosis or mild factor to improve the pregnancy rate. There is again no information comparing the hormonal profile and follicular development after letrozole and CC in ovulatory women.

The aim of this study is to compare the hormonal profile after the use of LTZ and CC in anovulatory PCOS women and ovulatory women with unexplained subfertility. The hypothesis is that the FSH risk after LTZ is shorter than that of CC.

ELIGIBILITY:
Inclusion criteria:

* Age of women 18-39 years
* Irregular menstrual cycles with anovulation (cycle >35 days) together with polycystic ovaries on pelvic scanning or laboratory/clinical hyperandrogenism (in PCOS group)
* Regular cycle of 25-35 days cycle for the ovulatory women group
* Body mass index </= 30 kg/m2

Exclusion criteria:

* Couples undergoing ART treatment cycles
* History of ovarian surgery
* Drug allergy to CC or LTZ
* History of diabetes mellitus or other severe medical diseases
* Refusal to join the study

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
FSH concentrations | Alternative day during ovulation induction cycle (for about 3 month)

SECONDARY OUTCOMES:
LHconcentration | Alternative day during ovulation induction cycles (for about 3 month)
Endometrial Thickness | Monitoring during ovulation induction cycle (for about 3 month)
Oestradiol concentration | Alternative day during ovulation induction cycles (for about 3 month)
Progesterone concentration | Alternative day during ovulation induction cycles (for about 3 month)
Number of growing follicles | Monitoring during OI cycles (for about 3 month)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Lee, MBBS, MRCOG, Principal Investigator — Queen Mary Hospital / University of Hong Kong.
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong